CLINICAL TRIAL: NCT04115605
Title: A 3 Years Naturalistic Cohort Survey of Altis Single Incision Sling System For Female Stress Urinary Incontinence A Post-marketing and Multicenter Prospective Observational Cohort Study in Subjects With Female Stress Urinary Incontinence
Brief Title: A 3 Years Naturalistic Cohort Survey of Altis Single Incision Sling System For Female Stress Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: SU017
Record Dates: First submitted 2015-07-23; First posted 2019-10-04 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Urinary Incontinence, Stress
Keywords: Single Incision Sling
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Altis Single Incision Sling — Minimally invasive system including permanently implantable synthetic suburethral sling for the surgical treatment of female Stress Urinary Incontinence

SUMMARY:
The purpose of this study is to monitor the use of Altis Single Incision Sling (SIS) in a real world population and collect medical data on effectiveness and to monitor safety of Altis SIS at 12 and 36 months post device implantation in women with stress urinary incontinence.

DETAILED DESCRIPTION:
This project has been launched after the introduction of Altis in Europe. This study is a multicenter prospective, observational (i.e. naturalistic) post-marketing clinical follow-up of women for who stress urinary incontinence was diagnosed and will be treated with Altis Single Incision Sling System. Therefore these patients will be asked to allow to use their clinical data and answer some questionnaires. The patients'data will be collected in routine clinical practice before, during and after surgery until 12 months. Then, questionnaires will be mailed to the participants annually during 2 additional years.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with Altis Single Incision Sling System

Exclusion Criteria:

* Refuses to be included in the survey or that their medical data will be used for research purposes
* Indication for Altis Single Incision Sling System implantation is not for the treatment of female urinary incontinence.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female implanted with Altis Single Incision Sling System to treat stress urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2023-09-22 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | 12 months
  PGI-I is a validated question that collects the patient's impression of improvement after the surgery. Among this 7 point-scale (very much better, much better, a little better, no change, a little worse, much worse and very much worse), the patients are asked to check the one number that describes how their urinay tract condition is now, compared with how it's was before the surgery. Patients who score little or much or very much better without serious or severe related adverse events will be considered a treatment success. The percentage of patients who describe the treatment success is measured
Adverse events | 12 months
  Adverse events are any toward medical occurrence, unintended disease or injury or any untoward clinical signs in subjects. Adverse events will be categorized according to relatedness to device or procedure, severity and frequency. At 12-months, The percentage of patients without any device related severe or serious adverse events is measured.

SECONDARY OUTCOMES:
Cough stress test (CST) | Baseline, 8 weeks and 12 months
  CST provides the means for documenting stress urinary incontinence. CST is considered "positive" if any leakage is noted with cough or valsava. The percentage of patients with positive and negative test will be calculated at baseline, at the post-operative visit and at one year
Post-void residual (PVR) volume | Baseline, 8 weeks and 12 months
  PVR volume will be collected pre- and post implant procedure up to 12 months. If the PVR volume is considered normal by the physician after the procedure it is not necessary to collect these data at the subsequent follow-up visits.
Pad Use | Baseline, 8 weeks, 12, 24 and 36 months
  The number of pads used will be collected. Patients will be considered to be pad free if they report never wearing pads or wear pads just for a sense of security.
International Consultation on Incontinence Questionnaire (ICIQ-UI) | Baseline, 8 weeks, 12, 24 and 36 months
  The ICIQ-UI Short Form is a seft-administred questionnaire to evaluate the frequency, severity and impact on quality of life of urinary incontinence. Question 1 asked, "How often do you leak urine?" Subjects were instructed to select among "none" (0), "about once a week or less often" (1), "2 or 3 times a week" (2), "about once a day" (3), "several times a day" (4), and "all the time" (5). Question 2 asked, "How much urine do you usually leak (whether you wear protection or not)?" Patients responded with "none" (0), "a small amount" (2), "a moderate amount" (4) or "a large amount (6). Question 3 asked, "Overall, how much does leaking urine interfere with your everyday life?" Participants chose a number from 0 (not at all) to 10 (a great deal). Question 1, 2 and 3 are summed to compute the total ICIQ score.The total score range is then a minimum of 0 to a maximum of 21. The mean score, aboslute and relative change compared to baseline will be measure
Subject global satisfaction questionnaire | 8 weeks, 12, 24, 36 months
  This non-validated questionnaire provides additional information concerning patient satisfaction. This survey consists of two questions: Question 1 "how satisfied are you with your surgery?". Among 5 point-scale (very satisfied, satisfied, not satisfied-not dissatisfied, dissatisfied and very dissatified), patient check the one items that best describes the subject satisfaction. We measure the percentage the patients who very satisfied and satisfied. The patients answer the question "Do you recommend this operation to a friend?" by "yes" or "no". We measure the percentage of patients who answer "yes".
Incontinence quality of life questionnaire (I-QoL) | Baseline, 8 weeks, 12, 24, 36 months
  The Incontinence quality of life questionnaire (I-QoL) is a validated survey questionnaire with 22 items that are scored on a 5-point Likert scale. The I-QOL ans its subcale scores are computed by adding each item's reponse, subtracting the lowest possible score and diving that sum by the possible raw score range. The scores are then transformed to have a range from 0 (maximum problem) to 100 (no problem at all). The mean score, absolute and relative change compared to baseline
Impact on sexual function assessed by the Pelvic organ/urinary incontinence sexual questionnaire (PISQ 12) | Baseline, 8 weeks, 12, 24, 36 months
  The Pelvic organ/urinary incontinence sexual questionnaire (PISQ-12) is a validated and reliable short form questionnaire including 12 questions that evaluates sexual function in heterosexual women with urinary incontinence and/or pelvic oragn prolapse. Reponses are graded on a 5-point Likert scale from "never" to "always". The scores will be calculated at each assessment visit. The mean score, absolute and relative change compared to baseline
Patient Global Impression of Improvement (PGI-I) | 8 weeks, 24, 36 months
  PGI-I is a validated question that collects the patient's impression of improvement after the surgery. Among this 7 point-scale (very much better, much better, a little better, no change, a little worse, much worse and very much worse), the patients are asked to check the one number that describes how their urinay tract condition is now, compared with how it's was before the surgery. The percentage of patients who describe very much better or much better or little better is measured
Adverse events | 8 weeks, 24, 36 months
  Adverse events are any toward medical occurrence, unintended disease or injury or any untoward clinical signs in subjects. Adverse events will be categorized according to relatedness to device or procedure, severity and frequency. The percentage of patients without any device related severe or serious adverse events is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Capon, MD, Principal Investigator — CHU Pellegrin, Bordeaux, France
Locations (33):
- UZ Leuven, Leuven, Belgium
- France (24):
  - CHRU Hotel Dieu, Angers
  - Clinique Rhône Durance, Avignon
  - Clinique Champeau Mediterranée, Béziers
  - CHU Pellegrin-Urology Departement, Bordeaux
  - CHU Pellegrin_Gyneacology Departement, Bordeaux
  - Polyclinique Jean Villars, Bruges
  - Hôpital du Pays d'Autan, Castres
  - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Victor Jousselin, Dreux
  - CH Paul Ardier, Issoire
  - Clinique Saint-Charles, La Roche-sur-Yon
  - Centre Hospitalier Saint Louis, La Rochelle
  - Clinique du Mail La Rochelle, La Rochelle
  - Clinique Saint-Amé, Lambres-lez-Douai
  - CH Libourne, Libourne
  - Clinique Mutualiste de la Porte de l'Orient, Lorient
  - Hôpital privé Jacques Cartier, Massy
  - Armand Brillart Hospital, Nogent-sur-Marne
  - CHI Poissy Saint Germain en Laye, Poissy
  - Clinique St Hilaire, Rouen
  - Centre Clinical, Soyaux
  - Clinique Saint Jean Languedoc, Toulouse
  - Clinique Ambroise Paré, Toulouse
- Germany (3):
  - Frauenärzte im Seenland, Gunzenhausen
  - Klinikum Memmingen, Memmingen
  - Klinikum Worms gGmbH, Worms
- Azienda USL Valle d'Aosta, Aosta, Italy
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Univeritario Joan XXIII, Tarragona
  - Hospital la Fé, Valencia
  - Hosital Clinico de Valladolid, Valladolid